CLINICAL TRIAL: NCT01563718
Title: VIVITROL® (Naltrexone for Extended Release Injectable Suspension (XR-NTX)) for Opioid Dependent Inmates Released From Prison
Brief Title: Pre-Release VIVITROL for Opioid Dependent Inmates
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIH VIVITROL -01; 3R01DA024549-03S1 (NIH)
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Naltrexone; vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRE-release XR-NTX (Experimental): Participants randomly assigned to the pre-release condition will receive one injection of XR-NTX 1-2 weeks prior to prison release plus up to five additional injections of XR-NTX in the community after release
  Interventions: Drug: naltrexone for extended release injectable suspension
- POST-release XR-NTX (Active Comparator): Participant randomly assigned to the post-release group will be referred to Rhode Island Hospital to receive up to six injections of XR-NTX immediately after release from prison
  Interventions: Drug: naltrexone for extended release injectable suspension

INTERVENTIONS:
Drug: naltrexone for extended release injectable suspension — VIVITROL (naltrexone for extended-release injectable suspension) is supplied as a microsphere formulation of naltrexone for suspension, at a dose of 4cc (380mg of naltrexone base), administered by intramuscular injection to the buttocks (alternating sides monthly) for six months.
  Other Names: VIVITROL

SUMMARY:
Naltrexone is a medication that has been shown to help prevent relapse to opioid addiction and it has been reported to be clinically effective in parolee populations although it is rarely used. Recently a depot formulation with one-month duration has received FDA approval for the treatment of alcoholism and opiate dependence. This means that rather than having to take medication daily, individuals can receive one injection that lasts for approximately 30 days. The purpose of this study is to determine whether this monthly injection of naltrexone is practical and useful in the prevention of relapse to opioids and re-incarceration when administered to inmates prior to release from prison. The investigators will also monitor HIV risk behaviors to determine whether the intervention reduces risky behaviors associated with intravenous drug abuse and the spread of viruses such as HIV and hepatitis C. Volunteers will be randomized to receive an injection of depot naltrexone prior to release from prison or to contact study personnel in the community following release. Participants assigned to receive naltrexone in prison will receive 1 injection in prison, and 5 additional monthly injections for 5 months upon release. Participants assigned to contact study personnel upon release will receive all 6 injections in the community at RIH after their release from the ACI. Patients in both groups will be given identical follow up monthly for six months including measures of opiate use by self-report, and urine tests. An additional scheduled urine test will take place each month between monthly visits. There will also be a 12-month follow-up period for participants in both groups, which will consist of 2 visits, spaced 6 months apart, meaning that participants will be enrolled in the study for a total of about 18 months. All participants will be asked to complete brief questionnaires at follow-up visits to assess things such as services received, drug use, and depression.

ELIGIBILITY:
Inclusion Criteria:

1. Incarcerated adults with known release date.
2. Meet DSM-IV criteria for current (and/or prior to incarceration) opioid dependence.
3. Not interested in agonist (methadone, buprenorphine) treatment.
4. Currently opioid free by history ('detoxed'), with negative urine for all opioids and no sign of opiate withdrawal after IV (or IM if no available venous access) injection of 0.8 mg naloxone.
5. Good health by medical history, physical examination and laboratory tests.
6. Age older than 18.
7. Understands and signs a consent form.
8. Able to speak and understand English.
9. Females: not pregnant (urine hCG negative at baseline and prior to each injection), not planning conception; and planning appropriate contraception if sexually active.

Exclusion Criteria:

1. Current drug or alcohol dependence requiring long term residential treatment that would interfere with outpatient study participation. Dependence on substances that commonly co-occur with opioid dependence (e.g. cocaine, cannabis, alcohol) that do not rise to this level of severity will not be exclusionary in order to achieve a maximally representative sample.
2. Liver failure and/or liver function test levels greater than three times normal.
3. Pregnancy, lactation, or failure to use adequate contraceptive methods;
4. Active medical illness that might make participation hazardous, e.g. untreated hypertension, hepatitis with AST or ALT > 3 times upper limit of normal, unstable diabetes or heart disease. Adequately treated medical conditions are acceptable.
5. Untreated psychiatric disorder that might make participation hazardous, e.g. untreated psychosis, bipolar disorder with mania, significant suicide risk. Adequately treated psychiatric disorders and appropriate psychotropic medications would be allowed.
6. History of allergic reaction to naltrexone;
7. Current chronic pain diagnosis for which opioids are required for pain relief.
8. Obesity (BMI of 40 or greater) to reduce the likelihood of injection site reaction.
9. Known intolerance and/or hypersensitivity to naltrexone, carboxymethylcellulose, or polylactide-co-polymers (PLG) or any other components of the diluents.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2012-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Proportion of opioid-free days | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Friedmann, MD, MPH, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States